CLINICAL TRIAL: NCT01002157
Title: The Effects of Vitamin K2 Supplementation on the Progression of Coronary Artery Calcification
Acronym: VitaK-CAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: VitaK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEC09-2-075; NL27372.068.09
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Calcification; Vitamin K; Trial; Treatment
MeSH Terms: conditions — Coronary Artery Disease | interventions — menaquinone 7; Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin K2 supplementation (Experimental)
  Interventions: Dietary Supplement: Menaquinone-7 (Vitamin K2)
- Placebo control (Placebo Comparator)
  Interventions: Other: Placebo capsules

INTERVENTIONS:
Dietary Supplement: Menaquinone-7 (Vitamin K2) — Menaquinone-7 (Vitamin K2)
  Arms: Vitamin K2 supplementation
Other: Placebo capsules — Capsules containing no Menaquinone-7
  Arms: Placebo control

SUMMARY:
Both Coronary Artery Calcification (CAC)and its annual progression are a strong predictors of cardiovascular events. The development of arterial calcification results from imbalance between calcification promoting and inhibiting factors. An important inhibitor of calcification is Matrix Gla Protein (MGP): a protein present in the vascular wall where it is synthesized by Vascular Smooth Muscle Cells (VSMC). MGP requires Vitamin K-mediated carboxylation to function properly. Deficiency of Vitamin K has been demonstrated to cause arterial calcification and a diet containing large amounts of Vitamin K2 was associated with lower CAC and cardiovascular risk. In animal studies, active supplementation of Vitamin K2 caused regression of existing arterial calcification. Therefore, the aim of this randomized, double-blind, placebo-controlled clinical trial is to investigate whether daily supplementation of Vitamin K2 (Menaquinone-7) to patients with established CAC will lead to a decreased progression-rate of CAC after 24 months of follow-up in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Baseline Coronary Computed Tomographic Angiography (CCTA) of sufficient quality
* Baseline Agatston calciumscore 100 - 400

Exclusion Criteria:

* Baseline-scan of insufficient quality
* Heart rate greater than 70 beats per minute during first scan.(despite adequate treatment with metoprolol)
* Chronic or paroxysmal Atrial Fibrillation
* Presence or scheduled coronary revascularization procedure
* History of myocardial infarction or stroke.
* Presence of Diabetes Mellitus.
* Known kidney disease or a Glomerular Filtration Rate (GFR)MDRD < 60 ml/min/1.73m2
* Malignant disease (exception: treated basal-cell or squamous cell carcinoma).
* Use of Vitamin K antagonists.
* A life-expectancy < 2 years
* Pregnancy or wish to become pregnant in the near future.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-10; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Coronary Artery Calcification-score progression | 12 and 24 months

SECONDARY OUTCOMES:
Arterial Stiffness measured by Carotid-Femoral Pulse-Wave Velocity | 0, 12 and 24 months
Carotid Intima Media Thickness | 0, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Kroon, MD, PhD, Principal Investigator — Maastricht University Medical Center; Peter de Leeuw, MD, PhD, Study Chair — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands